CLINICAL TRIAL: NCT00763074
Title: Clinical Trial of Exercise and Diet in Type 2 Diabetic Women
Brief Title: Exercise and Diet in Type 2 Diabetic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eulji University Hospital (Other)
Responsible Party: Kyung Wan Min, Diabetes Center, Eulji University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obesity_2006_1
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-09

CONDITIONS: Insulin Sensitivity; Type 2 Diabetes
Keywords: Intra-Abdominal Fat; Adipokines; Exercise; Diet therapy
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Placebo Comparator): Conventional education of life style intervention for type 2 diabetes
  Interventions: Behavioral: Standard life style modification for type 2 diabetes
- Diet (Active Comparator): Dietary calorie restriction
  Interventions: Behavioral: Diet restriction
- Exercise (Active Comparator): Encourage to increase exercise amount: more than 60min's of exercise with moderate activity level two times per day
  Interventions: Behavioral: Exercise
- Diet and exercise (Active Comparator): Intervention for both of exercise and diet
  Interventions: Behavioral: Diet and exercise

INTERVENTIONS:
Behavioral: Standard life style modification for type 2 diabetes — Two session of education for exercise and diet.
  ----------- Exercise: 30min/day x 4/week Diet: ideal body weight x 30~35kcal/day
  Arms: Control
Behavioral: Diet restriction — Education for diet and exercise every 2 weeks
  ----------- Dietary calorie restriction: reduce their usual intake by -500kcal/day
  Arms: Diet
Behavioral: Exercise — Education for diet and exercise every 2 weeks
  ----------- Exercise: more than 60min/day of exercise with moderate activity level twice per day
  Arms: Exercise
Behavioral: Diet and exercise — Education for diet and exercise every 2 weeks
  ----------- Exercise education like as exercise group and diet education like as diet group
  Arms: Diet and exercise

SUMMARY:
The purpose of this study was to evaluate the effects of 12 weeks' increased daily physical activity versus diet restriction on regional fat distribution, insulin sensitivity and adipokines including retinol binding protein-4 (RBP-4), leptin, adiponectin, and a new marker, adiponectin to leptin ratio (AL ratio), in type 2 diabetic women.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patient
* BMI>23kg/m2
* Female

Exclusion Criteria:

* The patients with co-morbidity such as heart failure, chronic kidney disease or liver cirrhosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Wan Min, Professor, Principal Investigator — Eulji University